CLINICAL TRIAL: NCT00916825
Title: Impact of a Family-oriented Rehabilitation Programme for Mothers With Breast Cancer and Their Children - Quality of Life and Psychological Health of Mothers and Their Children
Brief Title: Impact of a Rehabilitation Programme for Mothers With Breast Cancer and Their Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: Dept. of Child and Adolescent Psychiatry, Philipps University Marburg (Other); Rexrodt von Fircks Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RvF01 - 135/07
Record Dates: First submitted 2009-06-09; First posted 2009-06-10 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2010-02

CONDITIONS: Breast Cancer
Keywords: breast cancer; quality of life; children of somatically ill parents; psychological adaptation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 3-week family oriented rehabprogramme (Experimental): waiting control group
  Interventions: Behavioral: rehabilitation programme "getting better together"

INTERVENTIONS:
Behavioral: rehabilitation programme "getting better together" — Mothers and their children (age 0-16) take part in a 3-week, family-oriented oncological rehabilitation programme which consists of medical, psychological and psychooncological treatments for mothers and children.

SUMMARY:
About 1/3 of newly diagnosed breast cancer patients are mothers of children who still live at home. They face additional challenges and stress, their children are also affected by the mother's illness. The oncological rehabilitation programme "getting better together" focuses on these special family needs. This waiting-control-group study examines the effectiveness of the intervention by accompanying the patients and their children over the course of a year and assessing their quality of life and psychological health.

DETAILED DESCRIPTION:
About 1/3 of newly diagnosed breast cancer patients are mothers of children who still live at home. They face additional challenges and stress, their children are also affected by the mother's illness. The oncological rehabilitation programme "getting better together", administered by the Rexrodt von Fircks Foundation and the Clinic Ostseedeich in Groemitz, Germany, focuses on these special family needs. This waiting-control-group-study, designed and executed at the Philipps University Marburg Medical Center, Department of Child and Adolescent Psychiatry, examines the effectiveness of the intervention by accompanying the patients and their children over the course of a year and assessing their quality of life and psychological health.

The primary outcome measure for mothers is the health related quality of life as assessed by the EORTC QLQ-C30 and BR-23; children's adaptation is assessed with the ILK (Inventory for the Assessment of Quality of Life of Children and Adolescents) as well as the Strengths and Difficulties Questionnaire (SDQ)

ELIGIBILITY:
Inclusion Criteria:

* participants of the rehabilitation programme "getting better together"
* mothers of children up to the age of 16
* have been diagnosed with and treated for breast cancer for the first time in their lives
* chemotherapy or radiation therapy ended no less than 6 weeks ago

Exclusion Criteria:

* metastases

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 801 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Mothers' and children's Quality of Life (EORTC OLQ-C30, QLQ-BR23; ILK) | 4 weeks before, at the beginning & post treatment, 3 and 12 months follow-up

SECONDARY OUTCOMES:
Children's psychological difficulties (SDQ) | 4 weeks before, at the beginning & post treatment, 3 and 12 months follow-up
Mothers' Depressive Symptoms (BDI) | 4 weeks before, at the beginning and post treatment, 3 and 12 months follow up
Mother's Life Satisfaction | 4 weeks before, at the beginning & post treatment, 3 and 12 months follow up
Mothers' and children's Treatment Satisfaction | Post Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fritz Mattejat, PhD, Study Director — Philipps University Marburg Medical Center, Dept. of Child and Adolescent Psychiatry; Katja J John, DP (MA), Principal Investigator — Philipps University Marburg Medical Center, Dept. of Child and Adolescent Psychiatry
Locations (1):
- Klinik Ostseedeich, Grömitz, Germany

REFERENCES:
- [Derived] John K, Becker K, Mattejat F. Impact of family-oriented rehabilitation and prevention: an inpatient program for mothers with breast cancer and their children. Psychooncology. 2013 Dec;22(12):2684-92. doi: 10.1002/pon.3329. Epub 2013 Jun 13. PMID 23760766
- See also: Study homepage — http://www.ggw-begleitstudie.de
- See also: The homepage of the foundation who initiated the oncological rehab-programme — http://www.rvfs.de